CLINICAL TRIAL: NCT06232785
Title: Application of Remifentanil Target Controlled Infusion Combined With Ibuprofen Injection in Gynecologic Endoscopic Surgery of Female Motion Sickness Patients
Brief Title: Gynecologic Endoscopic Surgery of Female Motion Sickness Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Second Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021/018
Record Dates: First submitted 2024-01-07; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Motion Sickness; Postoperative Nausea and Vomiting; Ibuprofen
MeSH Terms: conditions — Motion Sickness; Postoperative Nausea and Vomiting | interventions — Ibuprofen; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ibuprofen Group (Experimental): Participants received 0.8g ibuprofen intravenously 30 minutes before the end of the procedure
  Interventions: Drug: Ibuprofen
- Sufentanil Group (Placebo Comparator): Participants received 0.2ug/kg of sufentanil intravenously 30 minutes before the end of the procedure
  Interventions: Drug: sufentanil

INTERVENTIONS:
Drug: Ibuprofen — 0.8g intravenous injection 30min before the end of the operation
  Arms: Ibuprofen Group
Drug: sufentanil — 0.2ug/kg intravenous injection 30min before the end of the operation
  Arms: Sufentanil Group

SUMMARY:
The goal of this clinical trial is to compare the analgesic effect of sufentanil and ibuprofen and the incidence of vomiting, and to choose better postoperative analgesic drugs for motion sickness patients.in describe participant population. The main questions it aims to answer are:

* Whether this anesthesia method can meet the analgesic needs of gynecological laparoscopic surgery.
* Whether this anesthesia method can reduce the incidence of nausea and vomiting in patients with motion sickness after gynecological laparoscopic surgery.

Participants will use target-controlled infusion anesthesia combined with 0.8g ibuprofen injection.

Researchers will compare with use of target-controlled infusion combined with sufentanil to see if the incidence of nausea and vomiting is higher.

DETAILED DESCRIPTION:
Abstract: Objective: To compare the analgesic effect of sufentanil and ibuprofen and the incidence of vomiting, and to choose better postoperative analgesic drugs for motion sickness patients. Methods: Sixty-eight female patients aged between 18 and 60 years with motion sickness were selected for gynecologic endoscopic surgery under general anesthesia. Sixty-eight female patients were randomly divided into two groups, Group B (ibuprofen group) and Group S (sufentanil group), using a random number table method. The initial plasma target concentration of propofol was set at 4ug/ml and adjusted using the titration method. Once the patient lost consciousness, the target concentration of remifentanil was set at 4ng/ml and rocuronium at 0.6mg/kg, followed by endotracheal intubation three minutes later. During the operation, the plasma target concentration of propofol was maintained at 5ug/ml and remifentanil at 4ng/ml, with adjustments made based on stress reaction levels. General anesthesia was sustained through continuous administration of rocuronium at doses of 5 µg/kg/min. In Group B (ibuprofen group), intravenous administration of ibuprofen (0.8g) took place within half an hour before the end of surgery; in Group S (sufentanil group), intravenous injection of sufentanil (0.2ug/kg) occurred half an hour before completion of the operation, along with intravenous injection of dexamethasone (5mg) five minutes prior to anesthesia induction to prevent postoperative nausea and vomiting in both groups. The following data were collected: duration of operation, pneumoperitoneum time, extubation time, respiratory recovery time; Incidence of postoperative nausea and vomiting at different time intervals: Postanesthesia care unit residence period (T1), 0-3h after extubation (T2), 3-6h after extubation (T3), 6-12h after extubation (T4), 12-24h after extubation (T5); Visual analogue pain score : Postanesthesia care unit residence period (T1), 0-3h after extubation (T2), 3-6h after extubation (T3), 6-12h after extubation (T4), 12-24h after extubation (T5); Frequency of use of analgesics and antiemetic drugs; Incidence of adverse reactions within 24 hours after surgery; Postoperative satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years old;
2. Class I - II patients according to the American Society of Anesthesiologists classification;
3. Body mass index : 20-27kg/㎡;
4. non-life-threatening diseases of heart, lung, brain, liver, kidney and other important organs;
5. No recent use of sedatives, opioids, non-steroidal drugs such as ibuprofen, antiemetic drugs.
6. No history of digestive tract ulcer;
7. Motion sickness patients undergoing gynecological endoscopic surgery under general anesthesia.
8. Postoperative analgesia pump is not required.

Exclusion Criteria:

1. Low weight, poor general state;
2. general anesthesia drug allergy;
3. Long-term use of painkillers, antiemetic drugs, or use of opioids within 12 hours before surgery.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Comparison of postoperative nausea and vomiting between the two groups | From the end of surgery until 24 hours after surgery
  Incidence of postoperative nausea and vomiting at different time intervals: Pstanesthesia care unit residence period (T1), 0-3h after extubation (T2), 3-6h after extubation (T3), 6-12h after extubation (T4), 12-24h after extubation (T5); postoperative nausea and vomiting grading 24h after surgery: According to the severity of postoperative nausea and vomiting， postoperative nausea and vomiting was divided into 1-4 grades. Grade I: no nausea or vomiting; Grade II: mild nausea, abdominal discomfort, but no vomiting; Grade III: obvious vomiting, but no contents of the vomit; Grade IV: Severe vomiting with gastric juices and other contents. Postoperatively PONV is considered to occur in patients with grade II or higher
Visual Analogue Score scores in postoperative resting state of patients in two groups | From the end of surgery until 24 hours after surgery
  Visual analogue pain score : Pstanesthesia care unit residence period (T1), 0-3h after extubation (T2), 3-6h after extubation (T3), 6-12h after extubation (T4), 12-24h after extubation (T5)； Pain score 24h after operation: Pain Assessment Scale was used to evaluate the analgesic effect of the two groups. 0 doesn't hurt; 1 to 3 points - mild pain; 4 to 6 points - moderate pain; Score 7-10 - severe pain
Comparison of vomiting between the two groups | From the end of surgery until 24 hours after surgery
  Postoperative vomiting score 24 hours after surgery: Postoperative vomiting was divided into 0-3 points according to the degree of vomiting. 0 score: no vomiting; 1 point: vomiting 1-2 times; 2 points: vomiting 3 to 5 times; 3 marks: vomiting > 5 times

SECONDARY OUTCOMES:
Extubation time | One minute after surgery
  the time from cessation of propofol and remifentanil infusion at the end of surgery to withdrawal of tracheal catheter
Respiratory recovery time | One minute after surgery
  the time from the end of surgery when propofol and remifentanil infusion were stopped to the time when patients resumed breathing on their own
Occurrence of adverse reactions | Within 24 hours of extubation
  The incidence of postoperative adverse reactions such as dizziness, headache, agitation, respiratory depression and skin pruritus were compared between the two groups
Score of patient satisfaction | From the end of surgery until 24 hours after surgery
  Patient satisfaction score: 0: very satisfied, 1: average, 2: unsatisfactory. A score of more than 1 is considered poor satisfaction
Time of pneumoperitoneum | From the beginning to the end of the surgery
  Intraoperative condition
Time of operation | From the beginning to the end of the surgery
  Intraoperative condition
Volume of fluids and blood loss | From the beginning to the end of the surgery
  Intraoperative condition

CONTACTS AND LOCATIONS:
Overall Officials: dan Tian, Principal Investigator — 15526852169
Locations (1):
- Second Hospital of Jilin University, Changchun, Jilin, China